CLINICAL TRIAL: NCT03210779
Title: Effect of Probiotic Tablets and Topical Probiotic Oil (Lactobacillus. Reuteri) on Oral Wound Healing (Pilot Study)
Brief Title: Effect of Probiotics on Oral Wound Healing - Pilot Study
Acronym: PROWOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Svante Twetman, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-2430
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Wound
Keywords: oral wound healing; probiotics
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Cross-over pilot trial
Who Masked: Participant, Care Provider
Masking Description: Double Blind (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L.reuteri (Active Comparator): L. reuteri DSM 17938/ATCC PTA L. reuteri DSM 17938/ATCC PTA lozenges three times daily for 16 days + L. reuteri DSM 17938/ATCC PTA L. reuteri DSM 17938/ATCC PTA probiotic oil, topically, once daily for 8 days.
  Interventions: Dietary Supplement: L. reuteri DSM 17938/ATCC PTA
- Placebo (Placebo Comparator): Placebo lozenges three times daily for 16 days and placebo oil once daily for 8 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938/ATCC PTA — Ingestion of active lozenge twice daily for 16 days and topical application of active oil once daily for 8 days
  Arms: L.reuteri
Dietary Supplement: Placebo — Ingestion of inactive lozenge twice daily for 16 days application of inactive oil once daily for 8 days
  Arms: Placebo

SUMMARY:
This research will study the healing of standardized wounds created in the oral mucosa of volunteer participants during daily intake of tablets and topical application of oil containing the probiotic bacterium Lactobacillus reuteri. Our null hypothesis is that the consumption and topical application of probiotic supplements containing L. reuteri does not improve clinical healing of oral wounds in healthy participants when compared to controls.

DETAILED DESCRIPTION:
Intervention: after informed consent and baseline collection of clinical data (age,sex), the participants will be randomly assigned to one of the order of the treatments. As a run-in period, they will be given a supply of probiotic or placebo tablets enough for seven days. The participants are instructed to take two tablets daily (one in the morning and one in the evening, days 0-7) and are asked to refrain from any other foods or supplements containing probiotics. On day eight, the participant will attend to the clinics and a punch biopsy will be performed. Depending on the allocation group, probiotic or placebo oil will be supplied. The participant will be instructed to apply the oil locally on the wound with a plastic microbrush for 9 days every evening, and strongly reinforced to continue with the assigned tablets twice daily. The participant will attend the clinics on days two, five and eight post-wounding for follow-up photographies of wound healing. The first intervention period terminates with a wash-out period of four weeks, and then the second run-in an intervention period start following the same procedures.

The probiotic tablets and the probiotic oil (at the recommended dose) contain 2x10^8 CFU of Lactobacillus reuteri. Both the placebo tablets and oil are identical in size and composition but without the addition of the probiotic strains. The tablets and oil are packed in identical pots/bottles with color coding. The code will be kept from the investigators until the analysis are finished. Both the tablets and oil are provided by BIOGAIA AB.

Clinical procedures and sampling

All clinical procedures and sample collections will be conducted by a qualified and authorized dentist from the Institute of Odontology, Section for Cariology, Endodontics, Pediatric Dentistry and Clinical Genetics, Faculty of Health and Medical Sciences, University of Copenhagen. Collected samples (saliva, wound exudate and bacterial smear) will be stored in a freezer at -80 °C until all samples from all patients are gathered -for a maximum of six months. Running of all collected samples at the same time allows laboratory analyses to be carried out efficiently and avoids errors.

Punch biopsy: on day eight, a standardized circular wound of 3.5 mm diameter and approximately 1.5 mm deep will be created in the mucosa of the hard palate with aid of a biopsy punch. The biopsy is performed under aseptic conditions and local anesthesia using lidocaine 2% combined with epinephrine for local hemostasis. A scalpel is used to remove the surface epithelium and underlying superficial connective tissue, which will be discarded according to biosafety regulations from the Institute of Dentistry, University of Copenhagen. After wounding, the wound site will be photographed (blind-coded) with an intraoral camera, placing a standard-sized 6 mm diameter template around the wound as reference. The participant will attend to the dental clinics on days two, five and eight post-wounding to have a photograph of the wound taken by Ph.D student Gina Castiblanco. The wound-size on photographs will be measured by two raters and will be expressed as the ratio of the wound surface area relative to the standard label size with aid of software (Canvas 7, ACD Systems of America). The endpoint will be the percentage of initial wound size, measured at days two, five and eight post-wounding.

Saliva sampling: six samples of unstimulated whole saliva (UWS) fro m each subject will be collected (one at baseline, one right after the run-in period and one at the end of the intervention period). For USW collection, the participant will be sitting in a comfortable position with the head slightly bent. The participant is asked to keep the eyes open and make as few moves as possible, including swallowing. Then, he/she is asked to rinse the mouth in water and spit it out again. Thereafter, he/she is instructed to let saliva flow out of the mouth down a designated plastic cup for ten minutes. Aliquots of saliva (1.5 ml) will immediately be placed on ice and stored in a freezer at -80 °C until further analysis.

Collection of wound exudate: eight samples of wound exudate will be collected in total. The wound site will be dried with cotton pellets and periopaper strips (ProFlow, Amityville, NY, USA) will be gently pressed on the wound for 20 s. In case of blood contamination, the strip is discharged and the sampling is repeated after five min. The volume of exudate is recorded using a Peritron 8000 (Proflow) and expressed in µL. One strip holds approximately 0.1-0.4 µL of exudate. The strips are then transferred to plastic tubes and stored at -80 until further analysis.

Bacterial smear collection: four bacterial smears will be sampled. A sterile swab will be passed through the wound site, placed in a plastic tube and stored freezed at -80 °C until further analysis. The smears will be subjected to conventional microbial cultivation to detects the presence/absence and counts of bacterial species commonly associated with delayed wound healing (β-hemolytic streptococci and S. aureus).

Perception of pain and discomfort: a one-page logbook will be handed to the participants at the beginning of each run-in period so they can register the intake of tablets and their own perception of pain and discomfort according to a VAS-scale. The participant is also encouraged to register factors that could possibly influence the outcome (physical activity and number of alcoholic drinks). The participant will be asked to bring the filled logbook in the end of the intervention period.

Perceived stress and general health: in the end of the intervention period, the participant will be asked to fill the validated General Heath Questionnaire GHQ-12 (10) and the validated Perceived Stress Scale (11). These factors (self-perception of stress and general health) are known to be possible cofounders of wound healing outcomes.

Compliance: at the beginning of each intervention period, the participants will be provided with tablets enough for 16 days and oil for topical use enough for nine days application. Compliance will be checked through the participant´s completion of a logbook in which the daily intake of tablets and oil application is registered. For the last appointment, the participants will be asked to bring the remaining tablets and oil for counting/estimating.

Data analysis: all data will be processed with the open source statistics software "R" and controlled for normal distribution. Multivariate and univariate analysis of variance (MANOVAs and ANOVAs) will be used to assess within-subject change over time. A p-value less than 0.05 will be considered statistically significant. The obtained results will be published in an internationally recognized journal. If the results cannot be published in a journal, they will be available at the website of the University of the Odontology Institute. We make emphasis in that positive, negative and inconclusive results will be published.

Data management: all collected data will be treated in compliance with the Act on Processing of Personal Data and "The Health Law". At inclusion the participants will be assigned a unique number and a separate protocol without personal identification number. This study will not be reported to "Datatilsynet" as it is a private scientific health project

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (no chronic compromising illnesses)
* Healthy oral conditions
* Good level of oral hygiene

Exclusion Criteria:

* Adults over 50 years old
* Previous allergic reaction to local anesthetics
* Compromised oral mucosa
* Systemic diseases
* Obesity
* Alcoholism
* Smoking habit
* Pregnancy
* Antibiotic therapy within the last two months
* Active infection that needs treatment with antibiotics
* Systemic medications (glucocorticoid steroids, non-steroidal anti-inflammatory drugs -NSAIDS, chemotherapy, anticoagulant therapy) Contraceptives allowed.
* Thrombocytopenia or any of various inherited coagulopathies.
* Patients undergoing radiotherapy
* Inability to provide informed consent by means of physical or mental handicap

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of initial wound size area, measured in digital photographs | 8 days
  The reference value (100%) will be the area before intervention. The percentage is calculated with the second measure (photograph after the intervention)

SECONDARY OUTCOMES:
Levels of salivary oxytocin and salivary IL-10, in pg/ml | 8 days
  As measured with standardized immuno-assays (ELISA kits)
Levels of TNF-α and Interleukin 1β in the wound exudate | 8 days
  As measured with standardized immuno-assays (ELISA kits)
Numerical estimation of S. aureus and β-haemolitic streptococci (CFU/ml) | 8 days
  As measured from bacterial cultures obtained from wound smears

CONTACTS AND LOCATIONS:
Overall Officials: Svante Twetman, PhD, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erdman SE, Poutahidis T. Probiotic 'glow of health': it's more than skin deep. Benef Microbes. 2014 Jun 1;5(2):109-19. doi: 10.3920/BM2013.0042. PMID 24675231
- [Derived] Twetman S, Pedersen AML, Yucel-Lindberg T. Probiotic supplements containing Lactobacillus reuteri does not affect the levels of matrix metalloproteinases and interferons in oral wound healing. BMC Res Notes. 2018 Oct 25;11(1):759. doi: 10.1186/s13104-018-3873-9. PMID 30359300